CLINICAL TRIAL: NCT03592823
Title: Effect of Hydroxychloroquine on Atrial Fibrillation Recurrence After Radiofrequency Catheter Ablation in Patients With Atrial Fibrillation
Brief Title: Effect of Hydroxychloroquine on Atrial Fibrillation Recurrence
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AF-1
Record Dates: First submitted 2018-06-25; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): receiving radiofrequency ablation and anticoagulant therapy
- hydrochloroquine (Experimental): receiving radiofrequency ablation, anticoagulant therapy and hydrochloroquine treatment (200 mg,bidpo)
  Interventions: Drug: Hydroxychloroquine Sulfate 200 Mg Tablet

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 200 Mg Tablet — 200 mg, bidpo.
  Arms: hydrochloroquine

SUMMARY:
Atrial fibrillation is the most common arrhythmia in clinic. It can lead to heart failure or stroke, and has a high disability rate and mortality rate. At present, although radiofrequency ablation can cure atrial fibrillation, the success rate is only 50~70%, and has a high recurrence rate. In recent decades, no effective new antiarrhythmic drugs have been introduced, but there are side effects in long-term application of the existing antiarrhythmic drugs. Therefore, it is urgent to provide new and effective antiarrhythmic drugs.

Autophagy level of atrial myocytes in atrial fibrillation patients was significantly higher than that in sinus rhythm. Hydrochloroquine (HCQ) is a hydroxychloroquine sulfate composed of 4- amino quinoline compounds. As an effective inhibitor for autophagy, HCQ could effectively prevent the increased autophagy level of atrial myocytes in atrial fibrillation rabbits, prevent atrial effective refractory period (AERP) shortening, and decrease the rate and duration of atrial fibrillation.

At present, hydroxychloroquine is mainly used in the treatment of rheumatic immune system diseases and anti malaria. Because of its good safety and small side effects, HCQ has become an indispensable member of drugs in the combined treatment of rheumatoid arthritis and systemic lupus erythematosus patients. In recent years, studies have reported that hydroxychloroquine plays an important role in the prevention and treatment of cardiovascular diseases. Chloroquine could effectively shorten the action potential of atrial myocytes by blocking the inward rectifier potassium ion channel (Kir2.1) and reducing the inward potassium ion current Ik1. HCQ could also reduce 72% (P=0.002), and 70% for the risk of coronary heart disease, stroke, and transient ischemic disease. So the investigators speculate that HCQ may be a potential drug to block the occurrence of acute atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Successful radiofrequency ablation of atrial fibrillation within 24 hours

Exclusion Criteria:

* History of cerebrovascular disease: ischemic stroke, cerebral haemorrhage and transient ischemic attack.
* History of cardiovascular disease:unstable angina, myocardial infarction, coronary revascularization and congestive heart failure.
* History of renal impairment.
* History of Type I diabetes mellitus or Type II diabetes uncontrolled.
* History of liver impairment.
* History of alcoholism or drug abuse.
* Known severe skin rash or damage.
* Known retinal pigmentation and visual field defect.
* Allergy to any component of hydroxychloroquine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of atrial fibrillation after radiofrequency catheter ablation | up to 1 year
  Recurrence rate of atrial fibrillation after radiofrequency catheter ablation

SECONDARY OUTCOMES:
Side effects | up to 1 year
  Side effects including Eye diseases, skin damage, death, heart failure, malignant arrhythmia and stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Electrocardiograph, Harbin, Heilongjiang, China